CLINICAL TRIAL: NCT05411939
Title: Investigating the Impact of a Shared Decision-Making Tool on Patient Attitudes and Behaviors Regarding Treatment for Knee Osteoarthritis
Brief Title: Investigating the Impact of a Shared Decision-Making Tool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2000032637; No NIH funding (Other: 01.10.24)
Record Dates: First submitted 2022-06-06; First posted 2022-06-09 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Videotape Recording; Standard of Care

STUDY DESIGN:
Intervention Model Description: This is a randomized control trial in which participants will be assigned to one of two arms. Patients in the control arm of the study will watch a short video and then receive standard of care counseling with an orthopaedic surgeon. Patients in the treatment arm of the study will watch a short video and then receive standard of care counseling with an orthopaedic surgeon that includes discussion of the SDMT. All patients will complete pre- and post-visit surveys designed to measure the severity of their knee osteoarthritis and their willingness to proceed with different treatment modalities.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Patients in the control arm of the study will watch a short video and then receive standard of care counseling with an orthopaedic surgeon.
  Interventions: Other: Video; Other: Standard of Care
- Shared Decision-Making Tool (Experimental): Patients in the treatment arm of the study will watch a short video and then receive standard of care counseling with an orthopaedic surgeon that includes discussion of the shared decision-making tool.
  Interventions: Other: Shared Decision-Making Tool; Other: Video; Other: Standard of Care

INTERVENTIONS:
Other: Shared Decision-Making Tool — The Shared Decision-Making Tool (SDMT) is designed to provide a personalized, patient- centered framework for clinical discussions regarding treatment options for knee osteoarthritis. The tool functions through patient input of information such as pain severity and current symptoms, alongside other demographic information such as age, race, and comorbidities, to offer a series of outcomes to better illustrate how the patient's specific disease presentation will progress. Ultimately, using the SDMT may impact patient behavior if patients change their treatment preferences after utilizing the tool. This can empower them to seek additional support over time and maintain communication with their orthopedist to ensure they are on a healthier path.
  Arms: Shared Decision-Making Tool
Other: Video — Short video that describes knee osteoarthritis and possible treatment options.
Other: Standard of Care — Standard of care counseling for a patient presenting with knee osteoarthritis.

SUMMARY:
The purpose of this research study is to learn more about how the use of a Shared Decision-Making Tool (SDMT) will impact a patient's decision-making to pursue treatment for knee osteoarthritis.

DETAILED DESCRIPTION:
The main purpose of this study is to determine the impact of the SDMT on patient decision- making regarding various treatment modalities for knee osteoarthritis. If the SDMT is found to be beneficial, it can be implemented to help engage patients in their care and support more efficient implementation of treatment suggestions. This subsequently will improve patient's quality of life. Getting patients who have not taken advantage of preventive care or healthy lifestyles to change is paramount to making the medical experience in America more equal for all its citizens and reducing total societal costs. Building provider-patient communication tools that resonate with all stakeholders should inform patients as they work to make health decisions that reflect their individual beliefs.

ELIGIBILITY:
Inclusion Criteria:

* age 45-64
* mild to moderate knee pain consistent with a diagnosis of osteoarthritis

Exclusion Criteria:

* known inflammatory disease diagnosis (ex. Lupus, Sjogren, or rheumatoid arthritis, prior knee replacement, acute knee trauma)
* BMI over 45
* persons from vulnerable populations

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Change in Impact of the shared decision-making tool on a patient's willingness to seek treatment for knee osteoarthritis | Baseline, Immediately after intervention, and Week 4
  The primary objective is to assess the impact of the shared decision-making tool on a patient's decision to seek treatment for knee osteoarthritis. This will be assessed using a survey with a 5-point scale that asks several questions about a patient's willingness to pursue specific treatment options (1 = not at all willing, 5 = completely willing). The change over time is assessed to see if the intervention changes the patient's willingness to consider different treatment options. To assess change a baseline survey, a survey immediately after the intervention, and survey 4 weeks later will be collected. Change = (Week 4 - Baseline) and Change = (Immediately after intervention - Baseline) and Change = (Week 4 - Immediately after intervention).

SECONDARY OUTCOMES:
Change in Impact of SDMT on patient understanding | Baseline, Immediately after intervention, and Week 4
  This outcome is assessed using survey questions with a 5-point scale response option (1 = do not understand disease progression, 5 = completely understand disease progression). One survey question asks how well participants understand their disease progression. This is assessed over time to see if the SDMT impacts patient understanding. To assess change a baseline survey, a survey immediately after the intervention, and survey 4 weeks later will be collected. Change = (Week 4 - Baseline) and Change = (Immediately after intervention - Baseline) and Change = (Week 4 - Immediately after intervention).
Change in Impact of SDMT on decision-making | Baseline, Immediately after intervention, and Week 4
  This outcome is assessed through a survey question with a 5-point scale response option (1 = did not impact, 5 = completely impacted). This question asks specifically how the discussion (either standard of care or SDMT) impacts the participants decision to pursue treatment. To assess the change a baseline survey, a survey immediately after the intervention, and survey 4 weeks later will be collected. Change = (Week 4 - Baseline) and Change = (Immediately after intervention - Baseline) and Change = (Week 4 - Immediately after intervention).

CONTACTS AND LOCATIONS:
Overall Officials: Daniel H Wiznia, MD, Principal Investigator — Yale University
Locations (3):
- United States (3):
  - Yale Medicine Multispecialty, Guilford, Connecticut
  - Yale Ortho Milford, Milford, Connecticut
  - Yale Ortho, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: Yes
De-identified patient data will be available to other researchers who assist study preparation for publication.
Supporting Information: Study Protocol, ICF
Time Frame: De-identified data will be kept for 5 years after the data is collected.
Access Criteria: Researchers involved in the project will discuss access with the principal investigator.

REFERENCES:
- [Background] Hsu H, Siwiec RM. Knee Osteoarthritis. 2023 Jun 26. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK507884/ PMID 29939661
- [Background] Johnson CB. A Personalized Shared Decision-Making Tool for Osteoarthritis Management of the Knee. Orthop Nurs. 2021 Mar-Apr 01;40(2):64-70. doi: 10.1097/NOR.0000000000000739. PMID 33756532
- [Background] Katz JN, Arant KR, Loeser RF. Diagnosis and Treatment of Hip and Knee Osteoarthritis: A Review. JAMA. 2021 Feb 9;325(6):568-578. doi: 10.1001/jama.2020.22171. PMID 33560326
- [Background] Marcelin JR, Siraj DS, Victor R, Kotadia S, Maldonado YA. The Impact of Unconscious Bias in Healthcare: How to Recognize and Mitigate It. J Infect Dis. 2019 Aug 20;220(220 Suppl 2):S62-S73. doi: 10.1093/infdis/jiz214. PMID 31430386

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/39/NCT05411939/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/39/NCT05411939/ICF_001.pdf